CLINICAL TRIAL: NCT05035537
Title: Hemodynamic Optimization with Perioperative Gold Directed Therapy (PGDT) in Kidney Transplant
Brief Title: PGDT in Patients Undergoing Kidney Transplant
Acronym: PGDT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Cristiana Laici, MD, Principal Investigator, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: PGDT2017
Record Dates: First submitted 2021-08-29; First posted 2021-09-05 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Kidney Transplant; Complications
Keywords: Perioperative Goal Directed Therapy; Kidney Transplant

STUDY DESIGN:
Intervention Model Description: All patients who met eligibility criteria were randomised, using a computer generated randomization list, to either Group 1 (PGDT, intervention group) where minimally invasive continuous CI monitor (Edwards ClearSight) was used to guide a goal directed fluid administration protocol, and Group 2 (control) managed according to local and international best practice guidelines using standard hemodynamic monitoring.
Who Masked: Participant
Masking Description: The patients (individual participants) are prevented from having knowledge of the interventions assigned
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (PGDT) (Experimental): Group 1(PGDT, intervention group) where minimally invasive continuous CI monitor (Edwards ClearSight) was used to guide a goal directed fluid administration protocol
  Interventions: Procedure: PGDT
- Group 2 (control) (No Intervention): Group 2 (control) managed according to local and international best practice guidelines using standard hemodynamic monitoring

INTERVENTIONS:
Procedure: PGDT — The minimally invasive continuous CI monitor (Edwards ClearSight) was used to guide an optimization of preload with the use of algorithms based on fluids, inotropes and/or vasopressors to achieve a certain goal in medium arterial pressure (MAP), cardiac index (CI) and stroke volume variation (SVV)
  Arms: Group 1 (PGDT)

SUMMARY:
This study is a multicentric randomized controlled trial comparing two groups of patients undergoing single or dual kidney transplantation from deceased donors. To reduce perioperative complications optimal fluid management is essential in patients undergoing kidney transplantation. Heart rate, Medium Arterial Pressure (MAP), Central Venous Pressure (CVP), and urine output have been proposed in the literature to guide perioperative fluid therapy. These criteria are routinely applied in clinical practice; however these criteria have shown low sensitivity and poor predictive of postoperative complication, especially if used alone. The traditional approach in renal transplantation is the volume infusion guided whit CVP to the point of no further fluid responsiveness, but this can lead to excess fluid which can damage the endothelial glycocalyx and lead to organ failure for a fluid shift into the interstitial space.

As a way to reduce postoperative complications in surgical patients, in recent years, several studies have examined Perioperative Goal Directed Therapy (PGDT) as fluid administration guided by optimization of preload with the use of algorithms based on fluids, inotropes and/or vasopressors to achieve a certain goal in stroke volume (SV), cardiac index (CI), or oxygen delivery (DO2). However results regarding the potential role of PGDT cannot be considered definitive, because the various studies on the subject have not all conformed to the same methods and have not uniformly applied the same measurements, so their results regarding the potential role of PGDT cannot be considered definitive.

The aim of this work is to compare the effects of PGDT with conventional fluid therapy in patients undergoing kidney transplantation achievable through implementation of the non invasive monitoring.

DETAILED DESCRIPTION:
To reduce perioperative complications optimal fluid management is essential in patients undergoing kidney transplantation. Heart rate, Medium Arterial Pressure (MAP), Central Venous Pressure (CVP), and urine output have been proposed in the literature to guide perioperative fluid therapy. These criteria are routinely applied in clinical practice; however these criteria have shown low sensitivity and poor predictive of postoperative complication, especially if used alone. The traditional approach in renal transplantation is the volume infusion guided whit CVP to the point of no further fluid responsiveness, but this can lead to excess fluid which can damage the endothelial glycocalyx and lead to organ failure for a fluid shift into the interstitial space.

As a way to reduce postoperative complications in surgical patients, in recent years, several studies have examined Perioperative Goal Directed Therapy (PGDT) as fluid administration guided by optimization of preload with the use of algorithms based on fluids, inotropes and/or vasopressors to achieve a certain goal in stroke volume (SV), cardiac index (CI), or oxygen delivery (DO2). However results regarding the potential role of PGDT cannot be considered definitive, because the various studies on the subject have not all conformed to the same methods and have not uniformly applied the same measurements, so their results regarding the potential role of PGDT cannot be considered definitive.

The aim of this work is to compare the effects of PGDT with conventional fluid therapy in patients undergoing kidney transplantation achievable through implementation of the non invasive monitoring.

MATERIAL AND METHODS. This study is a multicentric randomized controlled trial comparing two groups of patients undergoing single or dual kidney transplantation from deceased donors. All patients who will meet eligibility criteria will be randomised, using a computer generated randomization list, to either Group 1 (PGDT, intervention group) where minimally invasive continuous CI monitor (Edwards ClearSight) will be used to guide a goal directed fluid administration protocol, and Group 2 (control) managed according to local and international best practice guidelines using standard hemodynamic monitoring.

STUDY DESIGN. The study protocol will be developed across the intraoperative and postoperative periods. In the intraoperative phase all standard monitored parameters such as EKG, SpO2 (oxygen saturation by pulse oximetry), airway pressure etc. will be the same for both groups. Where ClearSight minimally invasive monitoring will be used (Group 1), hemodynamic optimization goals will be as follows: CI ≥ 2.5 L/min/m2 and the SVV <10%. Sequential interventions used to reach the hemodynamic goals are regulated by a flow-chart provided in the study protocol. In Group 2 conventional static hemodynamic parameters (CVP, IBP) are evaluated to achieve an intraoperative MAP ≥ 70 mmHg with corrective actions (fluids, vasoactive agents) implemented according to the recommendations of good clinical practice and international guidelines. Both groups will receive standard induction immunosuppression according to our centre's practice as well as corticosteroid bolus (or two boluses if a dual kidney transplant was performed) before graft reperfusion. In the postoperative period all patients will be transferred to a dedicated post-surgical intensive care unit. The same standardized fluid therapy regimen will be adopted across both groups. Patient data will be prospectively collected, according to the study protocol, by designated personnel using a digital case report form.

SAMPLE SIZE CALCULATION AND STATISTICAL ANALYSIS. The investigators speculate that in order to detect a minimum reduction in the primary outcome of at least 18%, considering a power of 80% and a type I error of 5%, a total of 200 patients would be needed (100 per group). All results will be summarized in the text as means, unless differently stated each time with measures of variability expressed using mean and standard deviation. When reporting medians, measures of variability will be indicated as interquartile range, minimum value, and maximum value. Difference between population means will be obtained using the 2-sample t test; difference between population proportions will be obtained with the chi-square test and Fisher's exact test. Graft survival will be calculated from the date of kidney transplant to the date of last follow-up evaluation, graft loss, or patient death. P-values below or equal to 0.05 are considered as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years,
* first single- or dual-kidney transplant from a deceased donor,
* absence of atrial fibrillation or other severe arrythmia,
* ASA (American Society of Anesthesiologists) class III-IV,
* presence of written expression of consent.

Exclusion Criteria:

* patients receiving a retransplant,
* patients receiving a combined liver-kidney transplant,
* patients receiving a transplant from a living donor .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Hospital stay | Through study completion, an average of 6 months
  The primary study outcome was to investigate whether the adoption of a PGDT protocol would reduce overall hospital stay.

SECONDARY OUTCOMES:
Incidence of postoperative surgical and medical complications | Through study completion, an average of 6 months
  Secondary endpoint was the detection of any significant change in the incidence of postoperative surgical (Clavien-Dindo Classification≥ 3) and medical (pulmonary or cardiovascular) complications
Incidence of delayed graft function and graft loss | Through study completion, an average of 6 months
  Secondary endpoint was the detection of any significant change in the incidence of delayed graft function and graft loss
ICU stay | Through study completion, an average of 6 months
  Secondary endpoint was the detection of any significant change in the ICU length of stay

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Siniscalchi, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna, Italy
Locations (2):
- Italy (2):
  - SOD Anestesia e Rianimazione dei Trapianti e Chirurgia Maggiore, Azienda Ospedaliero-Universitaria Ospedali Riuniti Umberto I - GM Lancisi - G Salesi, Ancona, Ancona
  - Dipartimento di Anestesia e Rianimazione - Città della salute e della scienza, Torino, Torino, Torino

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Biancofiore G, Cecconi M, Rocca GD. A web-based Italian survey of current trends, habits and beliefs in hemodynamic monitoring and management. J Clin Monit Comput. 2015 Oct;29(5):635-42. doi: 10.1007/s10877-014-9646-7. Epub 2014 Dec 12. PMID 25500761
- [Background] Perilli V, Aceto P, Sacco T, Modesti C, Ciocchetti P, Vitale F, Russo A, Fasano G, Dottorelli A, Sollazzi L. Anaesthesiological strategies to improve outcome in liver transplantation recipients. Eur Rev Med Pharmacol Sci. 2016 Jul;20(15):3172-7. PMID 27466988
- [Background] Vincent JL, Rhodes A, Perel A, Martin GS, Della Rocca G, Vallet B, Pinsky MR, Hofer CK, Teboul JL, de Boode WP, Scolletta S, Vieillard-Baron A, De Backer D, Walley KR, Maggiorini M, Singer M. Clinical review: Update on hemodynamic monitoring--a consensus of 16. Crit Care. 2011 Aug 18;15(4):229. doi: 10.1186/cc10291. PMID 21884645
- [Background] Lobo SM, Rezende E, Knibel MF, Silva NB, Paramo JA, Nacul FE, Mendes CL, Assuncao M, Costa RC, Grion CC, Pinto SF, Mello PM, Maia MO, Duarte PA, Gutierrez F, Silva JM Jr, Lopes MR, Cordeiro JA, Mellot C. Early determinants of death due to multiple organ failure after noncardiac surgery in high-risk patients. Anesth Analg. 2011 Apr;112(4):877-83. doi: 10.1213/ANE.0b013e3181e2bf8e. Epub 2010 Jun 8. PMID 20530615
- [Background] Pearse RM, Harrison DA, James P, Watson D, Hinds C, Rhodes A, Grounds RM, Bennett ED. Identification and characterisation of the high-risk surgical population in the United Kingdom. Crit Care. 2006;10(3):R81. doi: 10.1186/cc4928. Epub 2006 Jun 2. PMID 16749940
- [Background] Jhanji S, Thomas B, Ely A, Watson D, Hinds CJ, Pearse RM. Mortality and utilisation of critical care resources amongst high-risk surgical patients in a large NHS trust. Anaesthesia. 2008 Jul;63(7):695-700. doi: 10.1111/j.1365-2044.2008.05560.x. Epub 2008 May 16. PMID 18489613
- [Background] Fischer MO, Fiant AL, Boutros M, Flais F, Filipov T, Debroczi S, Pasqualini L, Rhanem T, Gerard JL, Guittet L, Hanouz JL, Alves A, Parienti JJ; PANEX3 study group. Perioperative hemodynamic optimization using the photoplethysmography in colorectal surgery (the PANEX3 trial): study protocol for a randomized controlled trial. Trials. 2016 Mar 22;17:159. doi: 10.1186/s13063-016-1278-4. PMID 27004412
- [Background] Hamilton MA, Cecconi M, Rhodes A. A systematic review and meta-analysis on the use of preemptive hemodynamic intervention to improve postoperative outcomes in moderate and high-risk surgical patients. Anesth Analg. 2011 Jun;112(6):1392-402. doi: 10.1213/ANE.0b013e3181eeaae5. Epub 2010 Oct 21. PMID 20966436
- [Background] Gomez-Izquierdo JC, Feldman LS, Carli F, Baldini G. Meta-analysis of the effect of goal-directed therapy on bowel function after abdominal surgery. Br J Surg. 2015 May;102(6):577-89. doi: 10.1002/bjs.9747. Epub 2015 Mar 11. PMID 25759947
- [Background] Walsh SR, Tang T, Bass S, Gaunt ME. Doppler-guided intra-operative fluid management during major abdominal surgery: systematic review and meta-analysis. Int J Clin Pract. 2008 Mar;62(3):466-70. doi: 10.1111/j.1742-1241.2007.01516.x. Epub 2007 Nov 21. PMID 18031528
- [Background] Ameloot K, Palmers PJ, Malbrain ML. The accuracy of noninvasive cardiac output and pressure measurements with finger cuff: a concise review. Curr Opin Crit Care. 2015 Jun;21(3):232-9. doi: 10.1097/MCC.0000000000000198. PMID 25922896
- [Background] Scolletta S, Franchi F, Romagnoli S, Carla R, Donati A, Fabbri LP, Forfori F, Alonso-Inigo JM, Laviola S, Mangani V, Maj G, Martinelli G, Mirabella L, Morelli A, Persona P, Payen D; Pulse wave analysis Cardiac Output validation (PulseCOval) Group. Comparison Between Doppler-Echocardiography and Uncalibrated Pulse Contour Method for Cardiac Output Measurement: A Multicenter Observational Study. Crit Care Med. 2016 Jul;44(7):1370-9. doi: 10.1097/CCM.0000000000001663. PMID 27097293
- [Background] Sangkum L, Liu GL, Yu L, Yan H, Kaye AD, Liu H. Minimally invasive or noninvasive cardiac output measurement: an update. J Anesth. 2016 Jun;30(3):461-80. doi: 10.1007/s00540-016-2154-9. Epub 2016 Mar 9. PMID 26961819
- [Background] van der Spoel AG, Voogel AJ, Folkers A, Boer C, Bouwman RA. Comparison of noninvasive continuous arterial waveform analysis (Nexfin) with transthoracic Doppler echocardiography for monitoring of cardiac output. J Clin Anesth. 2012 Jun;24(4):304-9. doi: 10.1016/j.jclinane.2011.09.008. PMID 22608585
- [Background] Stover JF, Stocker R, Lenherr R, Neff TA, Cottini SR, Zoller B, Bechir M. Noninvasive cardiac output and blood pressure monitoring cannot replace an invasive monitoring system in critically ill patients. BMC Anesthesiol. 2009 Oct 12;9:6. doi: 10.1186/1471-2253-9-6. PMID 19821993